CLINICAL TRIAL: NCT04501978
Title: A Multicenter, Adaptive, Randomized, Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Hospitalized Patients With COVID-19
Brief Title: ACTIV-3: Therapeutics for Inpatients With COVID-19
Acronym: TICO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); University of Copenhagen (Other); Medical Research Council (Other Government); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); Prevention and Early Treatment of Acute Lung Injury (Other); Cardiothoracic Surgical Trials Network (Other); Eli Lilly and Company (Industry); Vir Biotechnology, Inc. (Industry); GlaxoSmithKline (Industry); Brii Biosciences Limited (Industry); AstraZeneca (Industry); Molecular Partners AG (Industry); Pfizer (Industry); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 014 / ACTIV-3
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Covid19
Keywords: COVID-19; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; ACTIV-3; ACTIV3
MeSH Terms: conditions — COVID-19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — bamlanivimab; remdesivir; sotrovimab; cilgavimab and tixagevimab drug combination; ensovibep; lufotrelvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACTIV-3 Drug plus SOC (Experimental): Participants in this study will be randomized to receive one of the ACTIV-3 drug treatments plus Standard of Care (SOC) or placebo plus SOC
  Interventions: Biological: LY3819253; Biological: Remdesivir; Biological: VIR-7831; Biological: BRII-196/BRII-198; Biological: AZD7442; Drug: MP0420; Drug: PF-07304814
- Placebo plus SOC (Placebo Comparator): The placebo arm may be pooled across more than one experimental arm if multiple investigational drugs are available to be tested at the same time. If it is not possible to use matching placebo over more than one experimental arm, additional placebo arms will be included in the study
  Interventions: Drug: Placebo; Biological: Remdesivir

INTERVENTIONS:
Biological: LY3819253 — Participants are no longer being randomized to this intervention.
  Arms: ACTIV-3 Drug plus SOC
Drug: Placebo — Commercially available 0.9% sodium chloride solution. Administered by IV infusion
  Arms: Placebo plus SOC
Biological: Remdesivir — Provided to all study participants as SOC unless contraindicated for an individual patient.
Biological: VIR-7831 — Participants are no longer being randomized to this intervention.
  Arms: ACTIV-3 Drug plus SOC
Biological: BRII-196/BRII-198 — Participants are no longer being randomized to this intervention.
  Arms: ACTIV-3 Drug plus SOC
Biological: AZD7442 — Participants are no longer being randomized to this intervention.
  Other Names: AZD8895 + AZD1061
  Arms: ACTIV-3 Drug plus SOC
Drug: MP0420 — Participants are no longer being randomized to this intervention.
  Other Names: ensovibep
  Arms: ACTIV-3 Drug plus SOC
Drug: PF-07304814 — 250 mg per day for 5 days. Administered as a constant rate intravenous infusion. Suspended: Participants are not currently being randomized to this intervention.
  Arms: ACTIV-3 Drug plus SOC

SUMMARY:
This study looks at the safety and effectiveness of different drugs in treating COVID-19 in people who have been hospitalized with the infection. Participants in the study will be treated with either a study drug plus current standard of care (SOC), or with placebo plus current SOC.

DETAILED DESCRIPTION:
This is a master protocol to evaluate the safety and efficacy of multiple investigational agents aimed at modifying the host immune response to SARS-CoV-2 infection, or directly enhancing viral control in order to limit disease progression.

The protocol is for a randomized, blinded, controlled platform study that allows investigational drugs to be added and dropped during the course of the study. This allows for efficient testing of new drugs against placebo and standard of care (SOC) treatment within the same study. When more than one drug is being tested at the same time, participants will be randomly allocated to treatments or placebo.

Randomization will be stratified by study site pharmacy and disease severity. There are 2 disease severity strata: Participants without organ failure (severity stratum 1); and participants with organ failure (severity stratum 2).

An independent Data and Safety Monitoring Board (DSMB) will regularly review interim analyses and summarize safety and efficacy outcomes. For investigational drugs with minimal pre-existing safety knowledge, the pace of enrollment with be initially restricted, and there will be an early review of safety data by the DSMB. For the study of each agent, at the outset of the trial, only participants in disease severity stratum 1 will be enrolled. This will continue until approximately 300 participants are enrolled and followed for 5 days. The exact number will vary according to the speed of enrollment and the timing of DSMB meetings. Prior to expanding enrollment to also include patients in disease severity stratum 2, safety will be evaluated and a pre-specified futility assessment by the DSMB will be carried out using 2 ordinal outcomes assessed at Day 5.

Both ordinal outcomes are used to assess futility because it is currently unclear whether the investigational agents under study will primarily influence non-pulmonary outcomes, for which risk is increased with SARS-CoV-2 infection, in part, through mechanisms that may be different from those that influence pulmonary outcomes.

For investigational agents passing this futility assessment, enrollment of participants will be expanded, seamlessly and without any data unblinding, to include participants in disease severity stratum 2 as well as those in disease severity stratum 1. Future interim analyses will be based on the primary endpoint of sustained recovery and will use pre-specified guidelines to determine early evidence of benefit, harm or futility for the investigational agent. Participants will be followed for 18 months following randomization.

The international trials within this protocol will be conducted in several hundred clinical sites. Participating sites are affiliated with networks funded by the United States National Institutes of Health (NIH) and the US Department of Veterans Affairs.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Positive test for COVID-19 and progressive disease suggestive of ongoing COVID-19 infection.
* Symptoms of COVID-19 for ≤ 12 days.
* Require admission to hospital for acute medical care (not for purely public health or quarantine purposes).

Exclusion Criteria:

* Patients who have received plasma from a person who recovered from COVID-19 or who have received neutralizing monoclonal antibodies at any time prior to hospitalization.
* Patients not willing to abstain from participation in other COVID-19 treatment trials until after Day 5 of the study. Co-enrollment in certain trials that compare recommended Standard of Care treatments may be allowed, based on the opinion of the study leadership team.
* Any condition which, in the opinion of the responsible investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments.
* Patients considered unable to participate in study procedures.
* Women of child-bearing potential who are not already pregnant at study entry and who are unwilling to acknowledge strong advice to abstain from sexual intercourse with men or practice appropriate contraception through 18 months of the study.
* Women of child-bearing potential who are unwilling to acknowledge the strong advice to abstain from sexual intercourse with men or practice appropriate contraception through 5 weeks of the study (PF-07304814 investigational agent).
* Pregnant women (PF-07304814 investigational agents).
* Nursing mothers (PF-07304814 investigational agents).
* Men who are unwilling to acknowledge the strong advice to abstain from sexual intercourse with women of child-bearing potential or to use barrier contraception through 18 months of the study.
* Men who are unwilling to acknowledge the strong advice to abstain from sexual intercourse with women of child-bearing potential or to use barrier contraception through 5 weeks of the study (PF-07304814 investigational agent).
* Presence at study enrollment of any of the following:

  1. stroke
  2. meningitis
  3. encephalitis
  4. myelitis
  5. myocardial ischemia
  6. myocarditis
  7. pericarditis
  8. symptomatic congestive heart failure
  9. arterial or deep venous thrombosis or pulmonary embolism
* Current or imminent requirement for any of the following:

  1. invasive mechanical ventilation
  2. ECMO (extracorporeal membrane oxygenation)
  3. Mechanical circulatory support
  4. vasopressor therapy
  5. commencement of renal replacement therapy at this admission (i.e. not patients on chronic renal replacement therapy).
* Participants with moderate to severe hepatic impairment (i.e. Child-Pugh class B or C) or acute liver failure (PF-07304814 investigational agent).
* Participants receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450 (CYP) 3A4 (PF-07304814 investigational agent).
* Patients will be excluded if taking drugs which have a narrow therapeutic window that are substrates of CYP3A4, including but not limited to: astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, pimozide, quinidine, sirolimus, tacrolimus, and terfenadine (PF-07304814 investigational agent).
* Patients with a history of deep vein thrombosis or pulmonary thrombotic embolism (Prior to initial futility assessment of PF-07304814 investigational agent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2753 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Time from randomization to sustained recovery | Up to Day 90
  Sustained recovery defined as being discharged from the index hospitalization, followed by being alive and home for 14 consecutive days prior to Day 90.

SECONDARY OUTCOMES:
All-cause mortality | Thru Day 90
Composite of time to sustained recovery and mortality | Thru Day 90
Days alive outside short-term acute care hospital | Up to Day 90
Pulmonary ordinal outcome | Days 1-7, 14 and 28
  Oxygen requirements measured by 7 categories (1 = least severe, 7 = most severe). The participant's highest (i.e. most severe) observed score is used.
Pulmonary+ ordinal outcome | Days 1-7
  Extrapulmonary complications and respiratory dysfunction measured by 7 categories (1= least severe, 7 = most severe). The participant's highest (i.e. most severe) observed score is used.
Incidence of clinical organ failure | Thru Day 28
Composite of death or serious clinical COVID-19 related events | Thru Day 90
Composite of cardiovascular events and thromboembolic events | Thru Day 90
Composite of grade 3 and 4 clinical adverse events, serious adverse events (SAEs) or death | Thru Days 5 and 28
Incidence of infusion reactions | Thru Day 0
Composite of SAEs or death | Thru 18 months
Change in SARS-CoV-2 neutralizing antibody levels | Baseline to Days 1, 3, 5, 28 and 90
Change in overall titers of antibodies | Baseline to Days 1, 3, 5, 28 and 90
Change in neutralizing antibody levels | Baseline to Days 1, 3, 5, 28 and 90
Incidence of home use of supplemental oxygen above pre-morbid oxygen use | 18 months
  Measured as: Alive at home and no use of continuous supplemental oxygen for an uninterrupted 14 day period
Incidence of no home use of supplemental oxygen above pre-morbid oxygen use | 14 days
  Measured as: Alive at home for an uninterrupted 14 day period and no use of continuous supplemental oxygen at end of 14 day time period.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Jens Lundgren, Principal Investigator — INSIGHT Copenhagen International Coordinating Centre, Rigshospitalet, University of Copenhagen; Prof. James Neaton, Study Chair — INSIGHT Statistical and Coordinating Centre, University of Minnesota
Locations (135):
- United States (98):
  - Banner University Medical Center Tucson (Site 206-004), 1625 N. Campbell Avenue, Tucson, Arizona
  - Southern Arizona VA Healthcare System (Site 074-009), 3601 S. 6th Ave., Tucson, Arizona
  - Velocity Chula Vista (Site 080-034), 752 Medical Center Ct., Ste. 304, Chula Vista, California
  - Community Regional Medical Center (Site 203-005), 2823 Fresno Street, Fresno, California
  - Velocity San Diego (Site 080-035), 5565 Grossmont Center Drive, Building 2, Suite 1, La Mesa, California
  - VA Loma Linda Healthcare System (Site 074-017), 11201 Benton Street, Loma Linda, California
  - VA Long Beach Healthcare System (Site 074-026), 5901 East 7th Street (09/151-M2), Long Beach, California
  - Keck Hospital of USC (Site 301-020), 1500 San Pablo Street, Los Angeles, California
  - Cedars-Sinai Medical Center (Site 208-002), 8700 Beverly Blvd., Los Angeles, California
  - Ronald Reagan UCLA Medical Center (Site 203-002), 757 Westwood Plaza, Los Angeles, California
  - Sacramento VA Medical Center (Site 074-023), 10535 Hospital Way, Mather, California
  - Hoag Memorial Hospital Presbyterian (Site 080-026), One Hoag Drive, Newport Beach, California
  - Palo Alto VAMC (Site 074-005), 3801 Miranda Avenue, Palo Alto, California
  - UC Davis Health (Site 203-004), 2315 Stockton Blvd., Sacramento, California
  - VA San Diego Healthcare System (Site 074-016), 3350 La Jolla Village Drive, San Diego, California
  - UCSF Medical Center at Mount Zion (Site 203-007), 1600 Divisadero St., San Francisco, California
  - San Francisco VAMC (Site 074-002), 4150 Clement St., San Francisco, California
  - UCSF Medical Center (Site 203-001), Moffitt-Long Hospital, 505 Parnassus Ave., San Francisco, California
  - Stanford University Hospital & Clinics (Site 203-003), 300 Pasteur Dr., Stanford, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Site 066-002), 1124 W. Carson Street, CDCRC Building, Torrance, California
  - University of Colorado Hospital (Site 204-001), 12605 E. 16th Avenue, Aurora, Colorado
  - Denver Public Health (Site 017-004), 660 Bannock St., MC2600 (Infectious Disease Clinic), Denver, Colorado
  - National Jewish Health / St. Joseph Hospital (Site 204-003), 1400 Jackson Street, Denver, Colorado
  - West Haven VA Medical Center (Site 025-007), 950 Campbell Avenue, West Haven, Connecticut
  - MedStar Georgetown University Hospital (Site 067-001), 3800 Reservoir Road NW, Washington D.C., District of Columbia
  - MedStar Health Research Institute (Site 009-021), MedStar Washington Hospital Center, 110 Irving St., NW., Washington D.C., District of Columbia
  - Washington DC VA Medical Center (Site 009-004), 50 Irving Street NW, Washington D.C., District of Columbia
  - Bay Pines VAMC (Site 074-004), 10000 Bay Pines Blvd., Bldg. 100, Room 5B-104, Bay Pines, Florida
  - Baycare Health System (Site 301-025), Morton Plant Hospital, 300 Pinellas Street, Clearwater, Florida
  - North Florida/South Georgia Veterans Health System (Site 074-011), 1601 SW. Archer Road, Gainesville, Florida
  - Memorial Healthcare System (Site 648-002), Memorial Regional Hospital, 3501 Johnson Street, Hollywood, Florida
  - Miami VAMC (Site 074-003), 1201 NW 16 Street, Miami, Florida
  - Hillsborough County Health Department, University of South Florida (Site 032-001), Tampa, Florida
  - Emory University (Site 301-008), The Emory Clinic, Bldg. A, Suite 2236, 1365 Clifton Rd., NE, Atlanta, Georgia
  - Lutheran Medical Group (Site 301-010), 7916 W. Jefferson Boulevard, Fort Wayne, Indiana
  - Cotton O'Neil Clinical Research Center (Site 080-030), Stormont Vail Health, 1500 SW 10th Avenue, Topeka, Kansas
  - University of Kentucky Hospital (Site 210-004), 1000 South Limestone St., Lexington, Kentucky
  - Ochsner Clinic Foundation (Site 301-015), 1514 Jefferson Highway, New Orleans, Louisiana
  - University of Maryland Medical Center (Site 301-019), 22 South Greene Street, Baltimore, Maryland
  - Massachusetts General Hospital (Site 202-002), 55 Fruit Street, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Site 202-001), 330 Brookline Ave., Boston, Massachusetts
  - Baystate Medical Center (Site 201-001), 759 Chestnut Street, Springfield, Massachusetts
  - University of Michigan (Site 205-001), 1500 East Medical Center Drive, Ann Arbor, Michigan
  - Henry Ford Health System, Henry Ford Hospital (Site 014-001), 2799 W. Grand Blvd., Detroit, Michigan
  - Minneapolis Heart Institute Foundation (Site 301-026), Abbott Northwestern Hospital, 920 E 28th St. #100, Minneapolis, Minnesota
  - Hennepin Healthcare (Site 027-001), 701 Park Avenue, Minneapolis, Minnesota
  - Minneapolis VA Health Care System (Site 105-001), 1 Veterans Drive, Bldg 70, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center (Site 112-001), 500 Harvard St. SE., Minneapolis, Minnesota
  - University of Mississippi Medical Center (Site 202-005), 2500 North State Street, Jackson, Mississippi
  - VA St. Louis Healthcare System (Site 074-027), 915 North Grand Blvd., Rm. C201, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center/Mary Hitchcock Memorial Hospital (Site 301-024), One Medical Center Drive, Lebanon, New Hampshire
  - Cooper University Hospital (Site 019-001), One Cooper Plaza, Camden, New Jersey
  - SUNY Downstate Medical Center (Site 033-001), 450 Clarkson Ave., Brooklyn, New York
  - Maimonides Medical Center (Site 033-002), 4802 10th Avenue, Brooklyn, New York
  - Ichan School of Medicine at Mount Sinai (Site 301-012), One Gustave L. Levy Place, Box 1620, New York, New York
  - Lincoln Medical Center (New York Health and Hospitals/Lincoln) (Site 003-016), 234 E. 149th Street, The Bronx, New York
  - Montefiore Medical Center Weiler Hospital (Site 206-003), 1825 Eastchester Road, The Bronx, New York
  - Montefiore Medical Center Moses Hospital (Site 206-001), 111 E. 210th Street, The Bronx, New York
  - Duke University Hospital (Site 301-006), 2301 Erwin Road, Durham, North Carolina
  - Wake Forest University Health Sciences (Site 210-001), Medical Center Blvd, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center (Site 207-003), 234 Goodman Ave., Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center (Site 108-001), 11100 Euclid Avenue, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital (Site 207-005), 18101 Lorain Avenue, Cleveland, Ohio
  - Cleveland Clinic Foundation (Site 207-001), 9500 Euclid Avenue, Cleveland, Ohio
  - Cleveland Clinic Marymount Hospital (Site 207-006), 12300 McCraken Road, Garfield Heights, Ohio
  - Oregon Health & Science University (Site 208-003), 3181 SW Sam Jackson Park Rd., Portland, Oregon
  - Portland VA Healthcare System (Site 074-024), 3710 SW. US Veterans Hospital Road, Portland, Oregon
  - UPMC Magee-Womens Hospital (Site 209-003), 300 Halket Street, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital (Site 209-001), 200 Lothrop Street, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital (Site 209-005), 5230 Centre Avenue, Pittsburgh, Pennsylvania
  - Rhode Island Hospital (Site 080-036), 593 Eddy Street, Providence, Rhode Island
  - The Miriam Hospital (Site 080-039), 164 Summit Ave., Providence, Rhode Island
  - VA Providence Healthcare System (Site 074-025), 830 Chalkstone Ave., Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center (Site 074-015), 109 Bee Street, Charleston, South Carolina
  - MUSC Research Nexus Clinic (Site 210-002), 96 Jonathan Lucas St., CSB 214, Charleston, South Carolina
  - MUSC Health Florence Medical Center (Site 210-006), 805 Pamplico Highway, Florence, South Carolina
  - VA TVHS Nashville Campus (Site 074-022), 1310 24th Avenue South, Nashville, Tennessee
  - Vanderbilt University Medical Center (Site 212-001), 1211 Medical Center Drive, Nashville, Tennessee
  - Hendrick Medical Center (Site 080-014), 1900 Pine Street, Abilene, Texas
  - CHRISTUS Spohn Shoreline Hospital (Site 080-001), 600 Elizabeth Street, Corpus Christi, Texas
  - Parkland Health and Hospital Systems (Site 084-002), 5200 Harry Hines Blvd, Dallas, Texas
  - UT Southwestern Medical Center (Site 084-001), 1936 Amelia Court, 2nd Floor, Dallas, Texas
  - Baylor, Scott and White Health (Site 301-003), Baylor University Medical Center, 3500 Gaston Ave., Dallas, Texas
  - Memorial Hermann Hospital (Site 203-006), 6411 Fannin Street, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center (MEDV AMC) (Site 074-006), 2002 Holcombe Blvd., Houston, Texas
  - Texas Heart Institute (Site 301-017), 6770 Bertner, MC4-266, Houston, Texas
  - CHRISTUS Good Shepherd Medical Center (Site 080-031), 700 E. Marshall Ave., Longview, Texas
  - Intermountain Medical Center (Site 211-001), 5121 South Cottonwood Street, Murray, Utah
  - University of Utah Hospital (Site 211-002), 419 Wakara Way, Suite 207, Salt Lake City, Utah
  - LDS Hospital (Site 211-004), 8th Ave. C Street, Salt Lake City, Utah
  - University of Virginia Health Systems (Site 301-021), 1215 Lee Street, Charlottesville, Virginia
  - Virginia Commonwealth University Health System (Site 210-005), 1250 East Marshall Street, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital (Site 080-018), 1906 Belleview Avenue, Roanoke, Virginia
  - Salem VA Medical Center (Site 074-014), 1970 Roanoke Blvd., Salem, Virginia
  - Harborview Medical Center (Site 208-001), 325 9th Avenue, Seattle, Washington
  - Swedish Hospital First Hill (Site 208-005), 747 Broadway, Seattle, Washington
  - University of Washington Medical Center - Montlake (Site 208-006), 1959 NE Pacific Street, Seattle, Washington
  - West Virginia University (Site 301-023), One Medical Center Drive, Morgantown, West Virginia
- Denmark (10):
  - Aalborg Hospital (Site 625-005), Hobrovej 18, Aalborg
  - Aarhus Universitetshospital, Skejby (Site 625-002), Department of Infectious Diseases, Palle Juul-Hensens Boulevard 99, Aarhus N
  - Bispebjerg Hospital (Site 625-013), Bispebjerg Bakke 23, Copenhagen
  - Righospitalet (Site 625-006), Blegdamsvej 9,, Copenhagen Ø
  - Herlev/Gentofte Hospital (Site 625-012), Medicinsk Afdeling, Herlev Ringvej 75, Herlev
  - Nordsjællands Hospital (Site 625-009), Dyrehavevej 29, Hillerød
  - Hvidovre University Hospital, Department of Infectious Diseases (Site 625-001), Kettegård allé 30, Hvidovre
  - Kolding Sygehus (Site 625-011), Medicinsk Afdeling, Sygehusvej 24, Kolding
  - Odense University Hospital (Site 625-004), Infektionsmedicinsk Forskningsenhed, J.B. Winsløwsgade 4, Odense
  - Zealand University Hospital, Roskilde (Site 625-010), Sygehusvej 10, Roskilde
- Greece (5):
  - Democritus University of Thrace (Site 635-021), University General Hospital of Alexandroupolis, Dragana, Alexandroupoli, Evros
  - Evangelismos COVID-19 Unit, (Site 635-020), 1st Dept. of Pulmonary and Critical Care Medicine, Evangelismos General Hospital, Dept., Ipsilantou 45-47, Athens
  - 1st Respiratory Medicine Dept., Athens University Medical School (Site 635-015), Athens Hospital for Diseases of the Chest "Sotiria Hospital", 152 Mesogeion Ave., Athens
  - 3rd Dept. of Medicine, Medical School, NKUA (Site 635-022), Sotiria General Hospital, 152 Mesogeion Ave., Athens
  - Attikon University General Hospital (Site 635-009), 4th Dept. of Internal Medicine, Medical School, National and Kapodistrian University of Athens, 1 Rimini St., Haidari, Athens
- Institute of Human Virology Nigeria (IHVN) (Site 612-601), Plot 252, Herbert Macaulay Way, Central Business District, Abuja, Nigeria
- Wojewódzki Szpital Zakazny (Site 625-302), Wolska 37, Warsaw, Poland
- Tan Tock Seng Hospital (Site 612-201), National Centre for Infectious Diseases (NCID), 11 Jalan Tan Tock Seng, Singapore, Singapore
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol (Site 626-003), Infectious Disease Unit, Second Floor, Building Maternal, Road Canyet s/n, Badalona, Barcelona
  - Hospital Universitari Arnau de Vilanova (Site 626-035), Av. Alcalde Rovira Roure 80, Lleida, Leida
  - Hospital Del Mar (Site 626-025), Paseo Maritimo 25-29, Barcelona
  - Hospital Universitari Vall d'Hebron (Site 626-033), Passeig de la Vall d'Hebron 119-129, Barcelona
  - Hospital Clínic de Barcelona (Site 626-004), Carrer de Villaroel 170, Barcelona
  - Hospital Universitario de Bellvitge (Site 626-034), Carrer de la Feixa Llarga, s/n, Barcelona
  - Hospital General Universitario Gregorio Marañón (Site 626-001), Dr. Esquerdo, 46, Madrid
  - Hospital Clínico San Carlos (Site 626-017), Enfermedades infecciosas, C/Martin Lagos CN, Madrid
  - UCICEC (Clinical Trial Unit) Hospital Universitario La Paz (Site 626-012), Paseo de la Castellana 261, 2a planta Hospital Maternal, Madrid
- University Hospital Zurich (Site 621-201), Department of Infectious Diseases and Hospital Epidemiology, Raemistrasse 100, Zurich, Canton of Zurich, Switzerland
- Uganda (6):
  - MRC/UVRI and LSHTM Uganda Research Unit (Site 634-601), Entebbe Regional Referral Hospital, Entebbe
  - Gulu Regional Referral Hospital (Site 634-603), Laroo Division, PO Box 160, Gulu
  - Makerere University Lung Institute (Site 634-604), New Mulago Hospital Complex, Mulago Hill, Kampala
  - St. Francis Hospital, Nsambya (Site 634-607), Nsambya Road Nsambya Hill, P.O. Box 7146, Kampala
  - Lira Regional Referral Hospital (Site 634-605), Lira
  - Masaka Regional Referral Hospital (Site 634-606), MRC/UVRI and LSHTM Uganda Research Unit, Plot 6 Circle Road, PO Box 556, Masaka
- United Kingdom (3):
  - Royal Victoria Infirmary (Site 634-007), Queen Victoria Road, Newcastle upon Tyne, Northumbria
  - Royal Free Hospital (Site 634-006), Pond Street, Hampstead, London
  - Guy's and St. Thomas' NHS Foundation Trust (Site 634-011), London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mourad A, Grandits GA, Siegel LK, Engen N, Barkauskas C, Eriobu N, Jain MK, Jensen TO, Ginde A, Higgs E, Knox DB, Kitonsa J, Kim K, Malin JJ, Rapti V, Price DA, Mena Lora AJ, Mathews G, Mylonakis E, Murray TA, Sandkovsky U, Paredes R, Ramachandruni S, Reilly C, Vock D, Williamson JC, Young BE, Self WH, Lundgren J, Holland TL; INSIGHT ACTIV-3/TICO Study Group and the STRIVE Network. Long-term outcomes of passive immunotherapy for COVID-19: a pooled analysis of a large multinational platform randomized clinical trial. Clin Microbiol Infect. 2025 Jun;31(6):1053-1060. doi: 10.1016/j.cmi.2025.02.002. Epub 2025 Feb 6. PMID 39922466
- [Derived] Jensen TO, Grandits GA, Jain MK, Murray TA, Grund B, Shaw-Saliba K, Matthay MA, Abassi M, Ardelt M, Baker JV, Chen P, Dewar RL, Goodman AL, Hatlen TJ, Highbarger HC, Holodniy M, Lallemand P, Laverdure S, Leshnower BG, Looney D, Moschopoulos CD, Mugerwa H, Murray DD, Mylonakis E, Nagy-Agren S, Rehman MT, Rupert A, Stevens RA, Turville S, Weintrob A, Wick K, Lundgren J, Ko ER; ACTIV-3/TICO Study Group. Effect of Neutralizing Monoclonal Antibody Treatment on Early Trajectories of Virologic and Immunologic Biomarkers in Patients Hospitalized With COVID-19. J Infect Dis. 2024 Mar 14;229(3):671-679. doi: 10.1093/infdis/jiad446. PMID 37948759
- [Derived] ACTIV-3/TICO Study Group; Barkauskas C, Mylonakis E, Poulakou G, Young BE, Vock DM, Siegel L, Engen N, Grandits G, Mosaly NR, Vekstein AM, Rogers R, Shehadeh F, Kaczynski M, Mylona EK, Syrigos KN, Rapti V, Lye DC, Hui DS, Leither L, Knowlton KU, Jain MK, Marines-Price R, Osuji A, Overcash JS, Kalomenidis I, Barmparessou Z, Waters M, Zepeda K, Chen P, Torbati S, Kiweewa F, Sebudde N, Almasri E, Hughes A, Bhagani SR, Rodger A, Sandkovsky U, Gottlieb RL, Nnakelu E, Trautner B, Menon V, Lutaakome J, Matthay M, Robinson P, Protopapas K, Koulouris N, Kimuli I, Baduashvili A, Braun DL, Gunthard HF, Ramachandruni S, Kidega R, Kim K, Hatlen TJ, Phillips AN, Murray DD, Jensen TO, Padilla ML, Accardi EX, Shaw-Saliba K, Dewar RL, Teitelbaum M, Natarajan V, Laverdure S, Highbarger HC, Rehman MT, Vogel S, Vallee D, Crew P, Atri N, Schechner AJ, Pett S, Hudson F, Badrock J, Touloumi G, Brown SM, Self WH, North CM, Ginde AA, Chang CC, Kelleher A, Nagy-Agren S, Vasudeva S, Looney D, Nguyen HH, Sanchez A, Weintrob AC, Grund B, Sharma S, Reilly CS, Paredes R, Bednarska A, Gerry NP, Babiker AG, Davey VJ, Gelijns AC, Higgs ES, Kan V, Matthews G, Thompson BT, Legenne P, Chandra R, Lane HC, Neaton JD, Lundgren JD. Efficacy and Safety of Ensovibep for Adults Hospitalized With COVID-19 : A Randomized Controlled Trial. Ann Intern Med. 2022 Sep;175(9):1266-1274. doi: 10.7326/M22-1503. Epub 2022 Aug 9. PMID 35939810
- [Derived] ACTIV-3-Therapeutics for Inpatients with COVID-19 (TICO) Study Group. Tixagevimab-cilgavimab for treatment of patients hospitalised with COVID-19: a randomised, double-blind, phase 3 trial. Lancet Respir Med. 2022 Oct;10(10):972-984. doi: 10.1016/S2213-2600(22)00215-6. Epub 2022 Jul 8. PMID 35817072
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Wick KD, Siegel L, Neaton JD, Oldmixon C, Lundgren J, Dewar RL, Lane HC, Thompson BT, Matthay MA; ACTIV-3/TICO study group. RAGE has potential pathogenetic and prognostic value in nonintubated hospitalized patients with COVID-19. JCI Insight. 2022 May 9;7(9):e157499. doi: 10.1172/jci.insight.157499. PMID 35298440
- [Derived] ACTIV-3/Therapeutics for Inpatients with COVID-19 (TICO) Study Group. Efficacy and safety of two neutralising monoclonal antibody therapies, sotrovimab and BRII-196 plus BRII-198, for adults hospitalised with COVID-19 (TICO): a randomised controlled trial. Lancet Infect Dis. 2022 May;22(5):622-635. doi: 10.1016/S1473-3099(21)00751-9. Epub 2021 Dec 23. PMID 34953520
- [Derived] ACTIV-3/TICO Bamlanivimab Study Group; Lundgren JD, Grund B, Barkauskas CE, Holland TL, Gottlieb RL, Sandkovsky U, Brown SM, Knowlton KU, Self WH, Files DC, Jain MK, Benfield T, Bowdish ME, Leshnower BG, Baker JV, Jensen JU, Gardner EM, Ginde AA, Harris ES, Johansen IS, Markowitz N, Matthay MA, Ostergaard L, Chang CC, Goodman AL, Chang W, Dewar RL, Gerry NP, Higgs ES, Highbarger H, Murray DD, Murray TA, Natarajan V, Paredes R, Parmar MKB, Phillips AN, Reilly C, Rupert AW, Sharma S, Shaw-Saliba K, Sherman BT, Teitelbaum M, Wentworth D, Cao H, Klekotka P, Babiker AG, Davey VJ, Gelijns AC, Kan VL, Polizzotto MN, Thompson BT, Lane HC, Neaton JD. Responses to a Neutralizing Monoclonal Antibody for Hospitalized Patients With COVID-19 According to Baseline Antibody and Antigen Levels : A Randomized Controlled Trial. Ann Intern Med. 2022 Feb;175(2):234-243. doi: 10.7326/M21-3507. Epub 2021 Dec 21. PMID 34928698
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] ACTIV-3/TICO LY-CoV555 Study Group; Lundgren JD, Grund B, Barkauskas CE, Holland TL, Gottlieb RL, Sandkovsky U, Brown SM, Knowlton KU, Self WH, Files DC, Jain MK, Benfield T, Bowdish ME, Leshnower BG, Baker JV, Jensen JU, Gardner EM, Ginde AA, Harris ES, Johansen IS, Markowitz N, Matthay MA, Ostergaard L, Chang CC, Davey VJ, Goodman A, Higgs ES, Murray DD, Murray TA, Paredes R, Parmar MKB, Phillips AN, Reilly C, Sharma S, Dewar RL, Teitelbaum M, Wentworth D, Cao H, Klekotka P, Babiker AG, Gelijns AC, Kan VL, Polizzotto MN, Thompson BT, Lane HC, Neaton JD. A Neutralizing Monoclonal Antibody for Hospitalized Patients with Covid-19. N Engl J Med. 2021 Mar 11;384(10):905-914. doi: 10.1056/NEJMoa2033130. Epub 2020 Dec 22. PMID 33356051
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CDC (Centers for Disease Control and Prevention): Coronavirus (COVID-19) website — https://www.cdc.gov/coronavirus/2019-nCoV/index.html
- See also: A Participant's Guide to Clinical Trials (NIAID) — https://www.niaid.nih.gov/clinical-trials/participant-guide
- See also: Find a Clinical Trial (NIAID) — https://www.niaid.nih.gov/clinical-trials/find-a-clinical-trial
- See also: Clinical Trials at NIAID — https://www.niaid.nih.gov/clinical-trials
- See also: National Institute for Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: WHO COVID-19 treatment guidelines — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/technical-guidance/patient-management

DOCUMENTS (1):
  • Informed Consent Form (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT04501978/ICF_000.pdf